CLINICAL TRIAL: NCT04779814
Title: A Non-interventional Study Describing the Healthcare Resource Utilisation and Clinical Outcomes Associated With LivaNova Vagus Nerve Stimulation Therapy in the UK.
Brief Title: Non-interventional Study Describing Healthcare Resource Utilisation and Clinical Outcomes Associated With VNS Therapy in UK.
Acronym: DANTE
Status: Active, not recruiting | Type: Observational
Sponsor: LivaNova (Industry)
Collaborators: OPEN VIE Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: LNE801
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
Keywords: VNS; DRE; drug resistant epilepsy; Vagus Nervus Stimulation; Healthcare Resource Utilization
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Cohort 1: Demipulse®/Aspire HC® (30 adult subjects)
- Cohort 2: Demipulse®/Aspire HC® (30 pediatric subjects)
- Cohort 3: Aspire SR® (30 adult subjects)
- Cohort 4: Aspire SR® (30 pediatric subjects)
- Cohort 5: SenTiva® (30 adult subjects)
- Cohort 6: SenTiva® (30 pediatric subjects)

SUMMARY:
This is a UK, multi-center, non-interventional study based on the use of health service administrative and medical records (paper-based and/or electronic, as applicable) along with the use of prospectively collected subject-reported outcomes on experience with use of VNS therapy using validated and bespoke self-completion questionnaires. Data for hospital resource utilisation will be extracted from the Hospital Episode Statistics (HES) database.

DETAILED DESCRIPTION:
Failure to control seizures in subjects with treatment resistant epilepsy can have a significant burden on the healthcare system. Vagus Nerve Stimulation (VNS) is an adjunctive treatment for patients with drug resistant epilepsy and is reported to reduce the frequency of seizures in adults and children. However, real-world data on healthcare resource utilization by patients with treatment-resistant epilepsy and their clinical outcomes prior to and post VNS device implantation in the UK are limited. The current study aims to describe the resource utilization and clinical outcomes prior to and following the implantation of different VNS devices (Demipulse®/Aspire HC®, Aspire SR® and SenTiva®) in subjects with drug resistant epilepsy

ELIGIBILITY:
Inclusion Criteria:

Living subjects who meet all of the following criteria will be considered for enrolment:

* Clinical diagnosis of drug resistant epilepsy
* Subjects who have had their first VNS device (Demipulse®/Aspire HC®, Aspire SR® and SenTiva®) implanted at least 18 months prior to their enrolment in the study data (with no change in generator, battery or lead).
* For SenTiva® and Aspire SR®, AutoStim was first activated within 1 month of implantation.
* For SenTiva®, scheduled dosing mode was activated within 1 month of implantation.
* Subjects must be able and willing to provide informed consent; subjects aged 7-12 years old and 13-15 years old will be provided with appropriate information and consent forms to explain the study in age appropriate language. These subjects will be asked to provide their assent to take part in the study, with consent provided by their parent/carer. Subjects under 7 years will be included in the study with consent from their parent/carer. For adult subjects (≥16 years) lacking the mental capacity to consent, advice about participation will be sought from an appropriate consultee, according to the Mental Capacity Act 2005.
* Adult and paediatric subjects (aged over 2.5 years at study enrolment) with available medical records for at least 12 months prior to VNS device implantation.

Exclusion Criteria:

* Subjects whose medical records are not available for review.
* Deceased subjects.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female adult (aged ≥16 years at VNS implantation) and paediatric (aged 1-15 years at VNS implantation) subjects with epilepsy who have had a VNS device Demipulse®/Aspire HC®, Aspire SR® or SenTiva® implanted will be involved in this study.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in hospital resource utilization | 12-month pre- implantation of VNS device to 18-month post-implantation of VNS device
  Description of change in hospital resource utilization from the 12-month period pre- to the 18-month period post-implantation of VNS device in subjects with drug resistant epilepsy.

SECONDARY OUTCOMES:
Change in Seizure information using ILAE classification | 12-month pre- implantation of VNS device to 6-month, to 12-month and to 18-month post-implantation of VNS device
  Onset and current classification and any prior classification of seizures will be described using ILAE classification
Initial titration period for each VNS device | 18-month period post-implantation of VNS device.
  Description of initial titration period for each VNS device
Characteristics and demographics of subjects at the time of implantation of VNS Therapy. | Implant procedure
  Description of characteristics and demographics of subjects at the time of implantation of VNS Therapy.
Change of AED treatments | Change from 12-month pre- implantation of VNS device to 18-month post-implantation of VNS device
  Assess the change in anti-epileptic drugs including dose change
Change in Seizure severity | Change from 12-month pre- implantation of VNS device to 6-month, to 12-month and to 18-month post-implantation of VNS device
  Change in Seizure severity; using measures such as rescue medication and/or time to recovery.
Change in Seizure frequency | Change from 12-month pre- implantation of VNS device to 6-month, to 12-month and to 18-month post-implantation of VNS device
  Change in Seizure frequency (by seizure type*, if available) and any changes in frequency.
Change in frequency of status epilepticus. | Change from 12-month pre- implantation of VNS device to 6-month, to 12-month and to 18-month post-implantation of VNS device
  Change in frequency of status epilepticus.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Carter, Principal Investigator — Bristol Royal Hospital for Children
Locations (5):
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Bristol Royal Hospital For Children, Bristol
  - The Walton Centre, Liverpool
  - Nottingham Children's Hospital, Nottingham
  - Oxford University Hospital NHSFT, Oxford